CLINICAL TRIAL: NCT02710344
Title: Automated Telehealth to Improve Psychiatric Self-Management and Community Tenure
Brief Title: Using Telehealth to Improve Psychiatric Symptom Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah Pratt, Assistant Professor in Psychiatry, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 28105; R01MH107625 (NIH)
Record Dates: First submitted 2016-03-10; First posted 2016-03-16 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual care at community mental health care provider
- Telehealth (Experimental): Usual care at community mental health care provider PLUS psychiatric telehealth program with remote monitoring.
  Interventions: Behavioral: Telehealth Program

INTERVENTIONS:
Behavioral: Telehealth Program — Psychiatric telehealth program, content assigned based on diagnosis, entry to study requires psychiatric instability defined as use of emergency/high cost psychiatric services.
  Arms: Telehealth

SUMMARY:
The overarching aim of this study is to evaluate whether telehealth leads to better mental health outcomes and decreased use of acute and crisis-based mental health care services by randomly assigning 300 people with serious mental illness (SMI) and psychiatric instability receiving services at 1 of 2 community mental health centers (CMHCs), each of which offers integrated behavioral and primary health care, to either Health Home Usual Care alone or telehealth plus Health Home Usual Care for 12 months, with assessments at baseline, 3, 6 and 12 months.

DETAILED DESCRIPTION:
The overarching aim of this study is to evaluate whether telehealth leads to better mental health outcomes and decreased use of acute and crisis-based mental health care services by randomly assigning 300 people with serious mental illness (SMI) and psychiatric instability receiving services at 1 of 2 community mental health centers (CMHCs), each of which offers integrated behavioral and primary health care, to either Health Home Usual Care alone or telehealth plus Health Home Usual Care for 12 months, with assessments at baseline, 3, 6 and 12 months.

This study will evaluate the effectiveness of an automated, algorithmically-driven, customizable telehealth platform that provides education, teaches illness self-management, prompts users to enact coping strategies, and monitors symptoms on a daily basis to remotely detect early warning signs among people with SMI, moving beyond the existing telehealth approaches (mainly educational websites and videoconferencing) for assessing and providing education and therapy to people with SMI.

This study has two specific aims. Aim 1 is to compare the effectiveness of telehealth with Health Home Usual Care by measuring improvements at 6 and 12 months in illness self-management, psychiatric symptoms, and health self-efficacy. Aim 2 is to compare the effectiveness of telehealth with Health Home Usual Care by comparing total cost of emergency room visits and hospital days during the 12 months prior to baseline to total costs of emergency room visits and hospital days during the 12 months after baseline.

This study will evaluate a widely used automated telehealth program that has been modified and upgraded by the research team to incorporate curriculum drawn from illness self-management interventions for SMI developed by the investigators (i.e., Integrated Illness Management and Recovery (I-IMR) and HOPES). Unlike other telehealth devices, it does not require an internet connection and is an efficient and innovative way to provide illness self-monitoring and self-management education. Responses are entered by the user and forwarded to a secure server via cellular signal. The telehealth specialist will access the server daily through a secure website using a username and password.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Chart DSM-V Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, post-traumatic stress disorder, or major depression and meet criteria for serious mental illness;
* Enrolled in treatment at site for at least 3 months;
* Psychiatric instability as indicated by 2 or more emergency room visits or hospitalizations in the past year, or multiple calls to the psychiatric crisis line within 3 months (10 or more);
* Expressed willingness to participate in a telehealth program;
* Must be able to read English.

Exclusion Criteria:

* Currently residing in a nursing home or group home;
* Terminal physical illness which is expected to result in death within one year;
* Primary diagnosis of dementia, co-morbid diagnosis of dementia, or significant cognitive impairment as indicated by a Mini Mental State Examination (MMSE) score <24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-09; Primary Completion 2020-03 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Total Cost of Emergency Room Visits and Hospital Days | Change in total cost of emergency room visits and hospital days during the 12 months prior to baseline compared to 12 months after baseline
  Cost of emergency room visits and hospital days

SECONDARY OUTCOMES:
Psychiatric symptom severity as assessed using the Brief Psychiatric Rating Scale | Change in psychiatric symptom severity as assessed using the Brief Psychiatric Rating Scale from baseline to 3, 6, and 12 months
  psychiatric symptom severity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Greater Nashua Mental Health Center, Nashua, New Hampshire
  - The Providence Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No